CLINICAL TRIAL: NCT00693563
Title: Scheduled Telephone Intervention for Individuals With Spinal Cord Injury and Their Families: A Randomized Controlled Trial
Brief Title: Scheduled Telephone Intervention for Individuals With Spinal Cord Injury and Their Families
Acronym: SCILink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeanne Hoffman (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jeanne Hoffman, Associate Professor, University of Washington
Organization: University of Washington (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 32148-G
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): The Control Group will receive usual care following discharge from the inpatient rehabilitation unit.
- Treatment Group (Experimental): Scheduled Telephone Intervention
  Interventions: Behavioral: Scheduled Telephone Intervention

INTERVENTIONS:
Behavioral: Scheduled Telephone Intervention — Participants and their significant others will be contacted by telephone within 24 to 48 hours after discharge and 10 additional times at weeks 1, 2, 4, 6, and months 2, 3, 4, 6, 8, and 10. The frequent early telephone contacts are meant to address early concerns that frequently arise after discharge are expected to last between 30 and 45 minutes. Later phone calls may be brief if no concerns are raised and are expected to address resource needs as well as ongoing questions that arise through the first year after injury. Content of each phone call will be dependent on issues raised by each individual participant and their significant other and/or follow-up on concerns raised in prior phone contacts rather than a specific structured interview.
  Arms: Treatment Group

SUMMARY:
The purpose of this study is to evaluate whether scheduled telephone intervention with individuals with spinal cord injury (SCI) and their caregivers in the first year following discharge from acute inpatient rehabilitation will reduce rehospitalizations and emergency room visits as well as improve adjustment to SCI.

DETAILED DESCRIPTION:
This project is a two-group randomized control trial. The control group will receive usual care given to all patients being discharged from acute inpatient rehabilitation following SCI. At 6 months and one year post injury an examiner blinded to group status will contact Control Group participants to collect outcome data.

The Telephone Intervention group (Treatment Group) will also receive their usual care following discharge and a welcome letter, which will include the same information as the Control Group, but also remind them of the up-coming telephone call schedule. Treatment Group participants and their significant others will be contacted by telephone within 24 to 48 hours after discharge and 10 additional times at weeks 1, 2, 4, 6, and months 2, 3, 4, 6, 8, and 10. The frequent early telephone contacts are meant to address early concerns that frequently arise after discharge are expected to last between 30 and 45 minutes. Later phone calls may be brief if no concerns are raised and are expected to address resource needs as well as ongoing questions that arise through the first year after injury. Content of each phone call will be dependent on issues raised by each individual participant and their significant other and/or follow-up on concerns raised in prior phone contacts rather than a specific structured interview. Treatment Group participants will also be contacted at 6 months and one year post injury by the examiner blinded to group status to collect outcome data.

ELIGIBILITY:
Inclusion Criteria:

* new traumatic SCI
* inpatient acute rehabilitation at the SCI system hospital
* residence in the catchment area at the time of injury

Exclusion Criteria:

* lack of a telephone
* non-English speaking
* severe psychiatric condition such as psychosis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2007-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Counts of rehospitalizations (frequency and duration), emergency department visits, and clinic visits to address medical complications | one year

SECONDARY OUTCOMES:
Composite of 4 measures to assess adjustment to SCI: Center for Epidemiologic Studies-Depression Scale (CES-D)79; Perceived Quality of Life (PQOL)80; Craig Handicap and Reporting Technique (CHART)81; Health-Promoting Lifestyle Profile II82 | one year

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bombardier, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- See also: Northwest Regional Spinal Cord Injury System — http://sci.washington.edu